CLINICAL TRIAL: NCT00707525
Title: Incidence of EmbyoO Aneuploidies in Natural Versus Stimulated Cycles in the Same Women.
Brief Title: Embryo Aneuploidies and Ovarian Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr. Elena Labarta, Instituto Valenciano de Infertilidad, Spain
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0607-C-M09-EL
Record Dates: First submitted 2008-06-30; First posted 2008-07-01 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Embryo Aneuploidies
Keywords: aneuploidies, natural cycle, stimulated cycle, preimplantation genetic diagnosis
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Natural cycle oocyte donation
- 2 (Active Comparator): Stimulated cycle oocyte donation.
  * Long protocol down-regulation with a GnRH agonist, starting on the midluteal phase of the previous cycle with leuprolide acetate (0.2mg/day).
  * Once evidence of downregulation is documented, leuprolide will be halved to 0.1 mg daily.
  * COH with be carried on with gonadotropins (150UI/day of rFSH and 75 UI/day of HP-hMG). The dose can be adjusted according to ovarian response as judged by ultrasound and by serum oestradiol (E 2 ) concentrations.
  Interventions: Procedure: Preimplantation Genetic Diagnosis

INTERVENTIONS:
Procedure: Preimplantation Genetic Diagnosis — Preimplantation Genetic Diagnosis (PGD) is performed on the embryos resulting from these natural and stimulated cycles.
  Arms: 2

SUMMARY:
There is a considerable concern about the effects of controlled ovarian hyperstimulation (COH) for In Vitro Fertilization- Embryo Transfer (IVF-ET) on embryo quality and on the incidence of chromosomal abnormalities in oocytes and embryos.

The main question remaining is if COH may increase the aneuploidies rate in young and healthy women. Therefore, the primary endpoint of the present study is to analyse the incidence of chromosomal abnormalities in this group of patients (oocyte donors), either in oocytes obtained after a natural cycle or in those retrieved after a COH cycle. To get rid of the male factor influence, donated sperm will be used.

ELIGIBILITY:
Donor Inclusion Criteria:

* 18 to 35 years old.
* BMI: 18-25Kg/m2
* Regular menstrual cycles
* Normal kariotype
* No previous controlled ovarian hyperstimulation (COH) treatments.

Donor Exclusion Criteria:

* Endometriosis
* Policystic ovarian syndrome
* Recurrent miscarriages.

Recipient Inclusion Criteria

* Aged until 45 years old
* No systemic diseases
* Following egg and sperm donation treatment.

Recipient exclusion criteria:

* Uterine disease (polyps, myomas, mullerian defects)
* Recurrent miscarriages.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Embryo aneuploidies | 2 cycles

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Valenciano de Infertilidad, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Labarta E, Bosch E, Alama P, Rubio C, Rodrigo L, Pellicer A. Moderate ovarian stimulation does not increase the incidence of human embryo chromosomal abnormalities in in vitro fertilization cycles. J Clin Endocrinol Metab. 2012 Oct;97(10):E1987-94. doi: 10.1210/jc.2012-1738. Epub 2012 Aug 3. PMID 22865900